CLINICAL TRIAL: NCT01620957
Title: Analyse de l'activité cérébrale intrinsèque Pendant le Coma et Lors du Retour à la Conscience
Brief Title: Longitudinal Study of the Default-mode Network Connectivity in Brain Injured Patients Recovering From Coma
Acronym: ACI-Coma
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: University Hospital, Toulouse (Other); Association des Traumatisés du Crane et de la Face, Paris, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: C11-55 Inserm; 2012-A00009-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-04-11; First posted 2012-06-15 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2021-08

CONDITIONS: Coma
Keywords: Default-mode network; Difussion tensor imaging; Cortical thickness; Coma; Vegetative state; Minimally conscious state; Neural correlate of consciousness
MeSH Terms: conditions — Coma; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coma patients

SUMMARY:
Several studies in healthy volunteers have suggested that the synchronized functional connectivity in the DMN (Deafult-Mode Network) would sustain the mental content at rest, and when required, a switch in the activity between the DMN and other networks involved in specific congnitive functions, would occur. This interaction permit to make the hypothesis, that baseline brain activity is likely to shape our ongoing " stream of consciousness " and could correlate with conscious perception. The investigators hypothesized that DMN connectivity strength would be related to the level of consciousness of brain-damaged patients. The investigators will follow severely brain-injured patient in coma. Clinical examination using standardized behavioural scales: FOUR score (Full Outline of UnResponsivess), Coma Recovery Scale-Revised); and brain imaging assessesments using MRI (functional and anatomical connectivity, cortical thickness) will be performed at: 3 to 30 (visit 1), and 60 (visit 2) days after insult. If patient recover a normal conscious state between 30 and 60 days, an additional clinical and brain imaging assessment will be performed to identify related changes in brain activity (visit 1*) Monitoring of vital parameters will be performed in patients by a senior anaesthesiologist throughout the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Brain-damaged patients in coma (trauma or anoxic origin).
* Male and female, ranging in age from 18 to 75 years.

Exclusion Criteria:

* Withdrawal of consent from the patients (or the persons having legal responsibility for them).
* Sedation or general anaesthesia during assessement period (< 24 hours).
* MRI contraindications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will analyse DMN functional and anatomical connectivity in severely brain-injured patients in coma and during the first two month following brain injury. All patients will be admitted from one of the four Critical Care Units of University Teaching Hospital of Toulouse, France.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change of DMN resting state fMRI connectivity between 1 and 2 month after severe brain injury | VISIT1 = coma state (an expected average of 3 to 30 days after brain injury), VISIT2 = recovery phase (an expected average of 30 to 60 days). Finally, in case of full recovery during the recovery phase an additional assessment will be performed (VISIT1*)
  To date, the functional significance of DMN resting state connectivity patterns remain unclear. We hypothesized that DMN connectivity strength would be related to the level of consciousness of non-communicative brain-damaged patients, as assessed by standardized behavioural scales (FOUR score, CRS-R). Furthermore, we expected that a disruption of functional connectivity in the DMN could predict brain-damaged patient's recovery.

SECONDARY OUTCOMES:
Compare functional and structural DMN connectivity between 1 and 2 month after severe brain injury | VISIT1 = coma state (an expected average of 3 to 30 days after brain injury), VISIT2 = recovery phase (an expected average of 30 to 60 days). Finally, in case of full recovery during the recovery phase an additional assessment will be performed (VISIT1*)
  Functional DMN connectivity will be investigated using probabilistic independent component analysis. Structural connectivity counterpart, will be assessed by diffusor tensor imaging and cortical thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Stein Silva, MD, PhD, Principal Investigator — Inserm, Department of Anesthesiology and Critical Care at the University Teaching Hospital of Toulouse, France; Kader Boulanouar, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Institut National de la Santé et de la Recherche Medicale, U825, Toulouse, Haute Garonne, France

REFERENCES:
- [Result] Peran P, Malagurski B, Nemmi F, Sarton B, Vinour H, Ferre F, Bounes F, Rousset D, Mrozeck S, Seguin T, Riu B, Minville V, Geeraerts T, Lotterie JA, Deboissezon X, Albucher JF, Fourcade O, Olivot JM, Naccache L, Silva S. Functional and Structural Integrity of Frontoparietal Connectivity in Traumatic and Anoxic Coma. Crit Care Med. 2020 Aug;48(8):e639-e647. doi: 10.1097/CCM.0000000000004406. PMID 32697504
- [Result] Rosazza C, Sattin D, Sebastiano DR, Minati L, Leonardi M, Silva S. Disruption of posteromedial large-scale neural communication predicts recovery from coma. Neurology. 2016 Jul 5;87(1):120-1. doi: 10.1212/WNL.0000000000002853. No abstract available. PMID 27378806